CLINICAL TRIAL: NCT00052494
Title: A Phase I Study Of STI 571 (Gleevec) In Combination With Cisplatin/Irinotecan In Patients With Extensive Stage Small Cell Lung Cancer
Brief Title: Combination Chemotherapy and Imatinib Mesylate in Treating Patients With Extensive-Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PMH-PHL-008; CDR0000258487 (Registry Identifier: PDQ (Physician Data Query)); NCI-5684
Record Dates: First submitted 2003-01-24; First posted 2003-01-27 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Lung Cancer
Keywords: extensive stage small cell lung cancer; recurrent small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma | interventions — Cisplatin; Imatinib Mesylate; Irinotecan

ARMS (1):
- STI-571 with cisplatin and irinotecan (Experimental)
  Interventions: Drug: cisplatin; Drug: imatinib mesylate; Drug: irinotecan hydrochloride

INTERVENTIONS:
Drug: cisplatin
Drug: imatinib mesylate
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop tumor cells from dividing so they stop growing or die. Imatinib mesylate may stop the growth of tumor cells by blocking the enzymes necessary for their growth. Combining more than one chemotherapy drug with imatinib mesylate may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combining cisplatin, irinotecan, and imatinib mesylate in treating patients who have extensive-stage small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of imatinib mesylate when administered with cisplatin and irinotecan in patients with extensive stage small cell lung cancer.
* Determine the recommended phase II dose of imatinib mesylate in patients treated with this regimen.
* Determine the response rate, median duration of response, progression-free survival, median survival, and overall survival of patients treated with this regimen.

OUTLINE: This is a multicenter, dose-escalation study of imatinib mesylate.

Patients receive cisplatin IV over 1 hour on day 1 and irinotecan IV over 60 minutes on days 1, 8, and 15. Treatment repeats every 28 days for a maximum of 4 courses. Patients also receive oral imatinib mesylate daily continually for one week prior to, during, and after chemotherapy in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of imatinib mesylate until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, additional patients are treated at the recommended phase II dose (one dose level below the MTD).

PROJECTED ACCRUAL: A total of 12-24 patients will be accrued for this study within 1-2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed extensive stage small cell lung cancer

  * Incurable but amenable to treatment with chemotherapy
  * c-kit positive by immunohistochemistry of original biopsy or other metastatic site
* At least one unidimensionally measurable lesion

  * > 20 mm by conventional techniques or > 10 mm by spiral CT scan
  * No prior radiotherapy to target measurable lesion(s), unless there is documented disease progression
* No known brain metastases

PATIENT CHARACTERISTICS:

Age

* Not specified

Performance status

* ECOG 0-1 OR
* Karnofsky 70-100%

Life expectancy

* More than 6 weeks

Hematopoietic

* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin normal
* AST and/or ALT ≤ 2.5 times upper limit of normal

Renal

* Creatinine normal OR
* Creatinine clearance ≥ 60 mL/min

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Gastrointestinal

* No concurrent untreated upper gastrointestinal bleeding that has not been fully investigated
* No gastrointestinal disease that would impair drug absorption

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception prior to, during, and for 3 months after study participation
* No history of ototoxicity
* No history of peripheral neuropathy
* No traumatic injury within the past 21 days
* No ongoing or active infection
* No other concurrent significant medical condition that would preclude study participation
* No concurrent psychiatric condition or social situation that would preclude study compliance
* No other malignancy within the past 5 years except treated nonmelanoma skin cancer, carcinoma in situ, or stage A prostate cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics
* No prior chemotherapy
* No other concurrent chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* More than 4 weeks since prior radiotherapy
* No prior radiotherapy to more than 25% of marrow

Surgery

* More than 3 weeks since prior major surgery
* No prior surgical procedure impairing absorption

Other

* No prior c-kit-targeted therapy
* No concurrent therapeutic dose of warfarin

  * Mini-dose warfarin for prophylaxis and low-molecular weight heparin allowed
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational agents
* No concurrent amifostine
* No other concurrent anticancer therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2003-04; Primary Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark D. Vincent, MD, Study Chair — London Health Sciences Centre
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada